CLINICAL TRIAL: NCT06502756
Title: Development, Feasibility, Acceptability, and Preliminary Effectiveness of a Digital Cognitive Behavioral Therapy for Hazardous Alcohol Drinking: A Single-Arm Pilot Study With Predictive Modeling in South Korea
Brief Title: Evaluating a Digital Cognitive Behavioral Therapy for Hazardous Alcohol Use: A Pilot Study in South Korea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, YOUNG-CHUL JUNG, Professor, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: WCTP-A-D-1; BT210029 (Other Grant/Funding Number: Seoul Metropolitan Government, South Korea)
Record Dates: First submitted 2024-07-02; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: High-risk Drinkers; Hazardous Alcohol Use
Keywords: digital intervention; mobile app; high-risk drinkers; hazardous alcohol use; secondary prevention; digital cognitive behavioral therapy; digital health

STUDY DESIGN:
Intervention Model Description: uncontrolled, single-arm, pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mobile application SOBER (digital cognitive behavioral therapy) (Experimental): Participants in this group will access to the mobile app SOBER for 4 weeks. Sober is designed to provide digitalized brief-intervention and cognitive CBT-based education for high-risk drinkers. Participants are expected to engage with the app, completing tasks such as self-monitoring (daily log function that instructs participants to record their alcohol consumption, along with changes in mood, appetite and sleep quality). The app will collect data on adherence, including diary completion rates and app login frequency. Participants were also provided with a smart watch to collect biometric data throughout the duration of the study.
  Interventions: Device: SOBER, mobile Application providing digital CBT

INTERVENTIONS:
Device: SOBER, mobile Application providing digital CBT — SOBER is a software application (Android) that delivers cognitive behavioral therapy (CBT) in a structured and interactive manner. It analyzes patterns in participants' lifestyles to identify problematic behaviors related to their alcohol consumption. By providing tailored guidance and support, the app aims to help individuals make sustainable changes, ultimately reducing hazardous drinking. This approach combines the principles of CBT with the convenience and accessibility of digital technology, offering a personalized experience to support the reduction of alcohol consumption.

SUMMARY:
The goal of this single arm pilot study is to investigate the feasibility, acceptability and preliminary effectiveness of the mobile app SOBER; for reducing and preventing hazardous alcohol drinking.

The main questions it aims to answer are:

* Feasibility: How well participants adhere to the app's lessons?
* Acceptability: Participants' satisfaction with and perceived usefulness of the app.
* Preliminary Effectiveness: The number of days participants remain abstinent.

Participants will:

* Use the mobile application SOBER, which delivers digital cognitive behavioral therapy, for four weeks.
* Wear a smartwatch to collect biometric data throughout the study.
* Visit the clinic three times: at baseline (V1), two weeks after the initial visit (V2), and four weeks after the initial visit (V3).
* Be evaluated using various questionnaires about their alcohol consumption, mood, and stress levels at each visit.
* Receive psychiatric consultation with a board-certified psychiatrist regarding their alcohol consumption, based on the data entered into the mobile app.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 19 and 65 years.
* Individuals classified as high-risk drinkers (hazardous drinking): Alcohol Use Disorder Identification Test (AUDIT) score of 8 or higher
* Individuals who have been admitted for treatment of alcohol use disorder no more than once.
* Individuals who are assessed to have completed detoxification treatment for alcohol.
* Individuals who own a smartphone and can independently use apps on the smartphone.
* Individuals who voluntarily agree to participate in this clinical study and have signed the consent form (or whose representative has signed the consent form).

Exclusion Criteria:

* individuals with active and progressive physical illnesses or a life expectancy of less than 6 months
* individuals with major psychiatric comorbidities such as schizophrenia, bipolar disorder, or major depressive disorder
* pregnant women or those planning to become pregnant during the study
* individuals who had participated in another clinical study within four weeks prior to the screening for this study

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-05-26 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Study completion rate | From enrollment to the end of treatment at 4 weeks
  The feasibility of the intervention was assessed based on the completion rates of the study
Adherence rate | From enrollment to the end of treatment at 4 weeks
  The adherence rate of educational sessions in the application
Preliminary Effectiveness | asked at baseline (V1), two weeks (V2), and four weeks (V3).
  days abstinent (%) in the past two weeks
Acceptability | In the end of treatment at 4 weeks
  assessed through participant satisfaction and perceived usefulness of the app, evaluated using a Likert-scale.
  Participants were asked to rate their satisfaction with the app on a scale from 0 (Not satisfied at all) to 5 (Very satisfied); and usefulness of the app from 0 (Not useful at all) to 5 (Very useful).

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | Administered at baseline (V1), two weeks (V2), and four weeks (V3).
  The PHQ-9 is a 9-item self-administered scale for assessing the severity of depression. Score Range: 0-27. : Higher scores indicate more severe depression. Scores of 10 or above suggest the need for treatment of depression.
Alcohol Use Disorders Identification Test (AUDIT) Score | Administered at baseline (V1), two weeks (V2), and four weeks (V3).
  The AUDIT is a 10-item questionnaire designed to assess alcohol consumption, drinking behaviors, and alcohol-related problems. Higher scores indicate more severe alcohol-related issues. A score of 8 or above suggests hazardous or harmful alcohol use. Score Range: 0-40
Generalized Anxiety Disorder 7-item Scale (GAD-7) | Administered at baseline (V1), two weeks (V2), and four weeks (V3).
  The GAD-7 is a 7-item self-report scale for identifying probable cases of generalized anxiety disorder and assessing its severity. Score Range: 0-21. Higher scores indicate more severe anxiety. Scores of 10 or above suggest the presence of generalized anxiety disorder.
Perceived Stress Scale (PSS) | Administered at baseline (V1), two weeks (V2), and four weeks (V3).
  The PSS is a 10-item questionnaire measuring the perception of stress. Score Range: 0-40. Higher scores indicate higher perceived stress levels. There are no specific cut-off scores; rather, scores indicate the relative level of stress perceived by the individual
Clinical Institute Withdrawal Assessment for Alcohol Scale (CIWA-Ar) | Administered at baseline (V1), two weeks (V2), and four weeks (V3).
  The CIWA-Ar is a 10-item scale used to assess the severity of alcohol withdrawal symptoms. Score Range: 0-67. Higher scores indicate more severe withdrawal symptoms. Scores of 10 or above indicate the need for medical intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Young-Chul Jung, Professor, MD, PhD, Principal Investigator — Department of Psychiatry, Yonsei University College of Medicine Severance Hospital, Yonsei University Health System
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No